CLINICAL TRIAL: NCT04697524
Title: Integrative Palliative Care/Psycho-Oncology Telehealth Group Medical Visits for Patients With Advanced Cancer: A Pilot Study
Brief Title: Integrative Palliative Care/Psycho-Oncology Telehealth Intervention in Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20806; NCI-2020-11397 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Advanced Malignant Solid Neoplasm; Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
Keywords: Telehealth; Palliative Care
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Telemedicine; Spermine Synthase; Referral and Consultation; Quality of Life; Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1: Supportive care (GMV) (Experimental): Participants will take a baseline assessment to collect socio-demographic information and complete a series of patient-reported outcome assessments (PROs) prior to their first group medical visit (GMV). The GMV intervention will take place over four weekly sessions conducted virtually. At the completion of all four weekly GMV sessions, participants will be asked to complete an exit survey. Participants in phase one will not be contacted or followed after the exit survey.
  Interventions: Behavioral: Support Group Therapy; Behavioral: Symptom Management Service (SMS) Consultation; Other: Quality of Life (QOL) Questionnaires; Other: Interview
- Phase 2: Refined GMV (Experimental): Up to three new cohorts of participants are recruited to assess the acceptability and feasibility of the refined intervention based on the results from the Phase 1 group
  Interventions: Behavioral: Support Group Therapy; Behavioral: Symptom Management Service (SMS) Consultation; Other: Quality of Life (QOL) Questionnaires; Other: Interview

INTERVENTIONS:
Behavioral: Support Group Therapy — Virtual group meetings
  Other Names: Virtual Visit; Telehealth
Behavioral: Symptom Management Service (SMS) Consultation — Virtual individual meetings with symptom management service (SMS) over 5 minutes
  Other Names: SMS; Virtual Visit
Other: Quality of Life (QOL) Questionnaires — Administered at each study visit
Other: Interview — Virtual exit interview at end of study
  Other Names: Virtual Visit

SUMMARY:
This trial investigates whether a joint and integrative approach to cancer care using palliative care and psycho-oncology is possible, and if it's beneficial to patients with cancer that has spread to other places on the body (advanced). The information gained from this study may help patients to learn about the medicinal and non-medicinal strategies to cope with their symptoms and side effects of their diagnosis and treatment while receiving peer support, in addition to standard individualized medical care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop and refine a joint Integrative Palliative Care/Psycho-oncology telehealth group medical visit (GMV) intervention based on feedback from an open pilot study with patient exit interviews.

II. To determine the feasibility and acceptability of the telehealth GMVs in a separate, single-arm pilot evaluation among patients with advanced cancer.

SECONDARY OBJECTIVE:

I. To estimate the preliminary efficacy of the GMVs among patients with advanced cancer.

EXPLORATORY OBJECTIVES:

I. To assess the financial viability of the GMVs. II. To measure the utilization of other supportive care services at Helen Diller Family Comprehensive Cancer Center (HDFCCC) and the Osher Center 3 months post-treatment.

III. To measure the University of California San Francisco (UCSF) healthcare utilization of participants 3 months post treatment.

OUTLINE:

PHASE I: The group-based intervention is developed, tested, and continuously refined based on participant feedback. Within 14 days of the first weekly group intervention, patients complete baseline questionnaires over 30-45 minutes about their sleep habits, pain management, anxiety/depression, and other symptoms. Patients then participate in a telehealth group medical intervention program over 2 hours weekly for up to 4 sessions where they review topics specific to managing fatigue and sleep habits, managing pain, managing emotional distress, and managing other symptoms and advanced care planning. During the weekly sessions, patients have the opportunity to meet with their symptom management service (SMS) provider in a separate virtual space for individual consultation over 5 minutes to discuss symptoms that they do not feel comfortable sharing in the larger group. The SMS provider may recommend specific interventions or resources for patients to discuss with their oncology, primary care, integrative medicine, psycho-oncology, or palliative care providers as appropriate. Patients also participate in an exit interview over 30 minutes to 1 hour.

PHASE II: Based on the feedback given in the first phase, three new cohorts of participants are recruited to assess the acceptability and feasibility of the refined intervention using similar procedures as in Phase I.

After completion of study, patients are followed up at 7 and 14 days, and then up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Carry a diagnosis of an advanced solid tumor cancer (locally advanced or metastatic, i.e., stage III or IV cancer)
* Be age >= 18 years
* Be able to speak and read English
* Be able to navigate websites, fill out forms on the web, communicate by email, and have regular access to the internet (assessed by participant self-report)
* Be capable of independently utilizing an online platform for telehealth group medical visits in a private setting (assessed by participant self-report)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Be able to understand a written informed consent document, and be willing to sign it

Exclusion Criteria:

* Have a cognitive or psychiatric condition prohibiting study consent or participation determined by co-principal investigators (PIs) or referring provider
* Be too medically unstable (or expected to become so during the study period) to participate in a telehealth group medical visit determined by co-PIs or referring providers
* Does not have insurance coverage for telehealth group medical visits
* Have extensive hearing loss such that ability to participate in the study would be impaired as determined by co-PIs or referring provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Develop Categories for intervention refinement (Phase 1) | Up to 3 months
  Qualitative methods to analyze participant feedback obtained during exit interviews and code notes from by the existing domains: session relevance, delivery mode, ease of participation, suggested changes. A thematic content analysis will be performed to determine themes based on patterns and responses in these categories. Two coders will then meet to discuss the themes and reach agreement on final categories used to refine intervention for Phase 2 participants.
Proportion of participants enrolled | 14 days
  The proportion of eligible and approached patients who consent to participate.
Retention rate | Up to 3 months
  The percentage of patients who complete pre and post-treatment questionnaires.
Adherence rate | Up to 3 months
  Percentage of patients who complete 2 or more sessions. Will use one-sample negative binomial probability and tests of binomial proportions to compare rates of feasibility to hypothesized values.
Number of participants deemed ineligible or refusing to participate | Up to 3 months
  Number of participants who are determined to be ineligible before 1st virtual visit or refusal to participate before 1st visit and during treatment.
Frequency of Participant Ineligibility Reason | Up to 14 days
  For potential study candidates who are ineligible, we will log reasons for ineligibility
Frequency of Participant Refusal Reason | Up to 14 days
  For potential study candidates who decide not to participate, we will log reasons for refusal.
Mean post-treatment participant satisfaction ratings | 1 day
  Participant ratings on intervention convenience, helpfulness, recommendation to others, worth doing, and feeling connected with University of California, San Francisco (UCSF). Descriptive statistics (frequencies, means, and standard deviations (SDs)) and 95% confidence intervals will summarize patients' ratings

SECONDARY OUTCOMES:
Change in distress score on the Edmonton Symptom Assessment System (ESAS) | Up to 3 months
  This 8-item questionnaire is used currently in the Symptom Management Service (SMS) and completed at each visit which measures severity at the time of assessment of each symptom and is rated from 0 to 10 on a numerical scale; with 0 meaning that the symptom is absent and 10 that it is the worst possible severity items (pain, activity, nausea, depression, anxiety, drowsiness, appetite, and sensation of well-being) . The sum of the scores for all symptoms is defined as the symptom distress score.
Change in scores on the Patient Health Questionnaire-8 (PHQ-8) | Up to 3 months
  The PHQ-8 is used to measure depression symptoms. The total Patient Health Questionnaire-8 (PHQ-8) score is calculated by combining the responses of the participant on questions addressing how bothered the participant has been by various problems over the past 2 weeks. Each of the 8 items is scored on a scale of 0 ("Not bothered at all") to 4 ("Nearly every day"). A total score of 0-4= No depression, 5-9='Mild Depression", 10-4="Moderate Depression", 15-19="Moderately severe depression", and 20 or higher ="Severe Depression".
Change in score on the Generalized Anxiety Disorder Assessment (GAD-7) | Up to 3 months
  The GAD-7 is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater
Change in score on the Patient Reported Outcomes Measurement Information System-Cancer (PROMIS) Pain Interference- Short Form 4a | Up to 3 months
  This 4-item questionnaire to measure the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities based on responses to statements about how the participants feel with a with a response ranging from 1="Never" to 5="Always", and a total raw score ranging from 4 - 20, which are converted to a scaled T-score (range 41.6 to 75.6) with higher scores indicating a greater hinderance to engagement in activities based on how much pain participants are experiencing.
Change in score on the PROMIS Sleep Disturbance- Short Form 6a | Up to 3 months
  This 6-item questionnaire to measure sleep disturbance based on responses to statements about how the participants feel with a response ranging from 1="Never" to 5="Always", and a total raw score ranging from 6 - 30, which are converted to a scaled T-score (range 31.7 to 73.3) with higher scores indicating a greater feeling of sleep disturbance.
Change in score on the PROMIS Fatigue - Short Form 6a | Up to 3 months
  This 6-item questionnaire to measure fatigue based on responses to statements about how the participants feel with a response ranging from 1="Never" to 5="Always", and a total raw score ranging from 6 - 30, which are converted to a scaled T-score (range 33.4 to 76.8) with higher scores indicating a greater feeling of fatigue.
Change in score on the PROMIS Social Isolation -Short Form 4a Short Form 4a | Up to 3 months
  This 4-item questionnaire to measure social isolation based on responses to statements about how the participants feel with a response ranging from 1="Never" to 5="Always", and a total score ranging from 4 - 20 which are converted to a scaled T-score (range 34.8 to 74.2) with higher scores indicating a greater feeling of social isolation.
Change in score on the Cancer Behavior Inventory-Brief (CBI-B) | Up to 3 months
  The Cancer Behavior Inventory-Brief Version (CBI-B), a 12-item measure of self-efficacy for coping with cancer. Participants rate each item on how confident they are that they can do that behavior. Responses range from 1 to 9 with 1="Not at all confident", 5="Moderately Confident" and 9="Totally confident". Numbers in the middle of these cut points indicate somewhat confidence in performing these behaviors to a lesser or greater degree but are not specifically labelled. The total score is calculated by summing the scores for the 12 items for a total score range of 12-98, with higher scores indicating greater coping efficacy.
Change in score on the Functional Assessment of Cancer Therapy- General (FACT-G) | Up to 3 months
  The FACT-G is a 27-item questionnaire designed to measure four domains of health related quality of life (HRQOL) in cancer patients with 4 domains of interest: Physical, social, emotional, and functional well-being. Each item response score ranges from 0 (not at all) to 5 (very much). The total score is a sum of the subscale scores, with a range from 0 - 108. The higher the score, the better the HRQOL.
Change in scores on the Quality of Life question | Up to 3 months
  This is a single-item question, "How would you rate your overall quality of life?" with responses ranging from a scale of 1 to 10 with greater scores indicating a greater quality of life. This is a validated measure used currently in the SMS.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cheng, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No